CLINICAL TRIAL: NCT02201030
Title: Multi-Center, Randomized, Double-Blind, Phase III Trial to Assess the Immunogenicity and Safety of Primary Vaccination With NBP606 in Healthy Infants
Brief Title: Immunogenicity and Safety Study of NBP606 in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NBP606_PCVI_III_2013
Record Dates: First submitted 2014-07-16; First posted 2014-07-25 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2016-10

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBP606 (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: NBP606
- Prevnar13 (Active Comparator): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: Prevnar13

INTERVENTIONS:
Biological: NBP606 — A single intramuscular injection into the thigh
  Arms: NBP606
Biological: Prevnar13 — A single intramuscular injection into the thigh
  Arms: Prevnar13

SUMMARY:
This study will assess the immunogenicity and safety of primary vaccination with NBP606 compared to the existing commercial vaccine, when given concomitantly with routine pediatric vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Infants between 42 and 98 days of age (approximately 2 months) at the time of enrollment.
* The LAR (Legally Authorized Representative) who understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

* Known hypersensitivity to any components of the pneumococcal vaccine
* Any confirmed or suspected immunosuppressive or immunodeficient conditions
* Coagulation disorder contraindicating IM(intramuscular) vaccination
* Subject has received any licensed vaccine(not including BCG and Hepatitis B)
* Participation to another study

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 577 (Actual)
Dates: Start 2014-09-06 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with the targeted antibody concentration | 1 month after the primary vaccination

SECONDARY OUTCOMES:
Geometric mean concentration ratio | 1 month after the primary vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Confidential Investigator, Principal Investigator — Clinical Research Center
Locations (1):
- Confidential, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided